CLINICAL TRIAL: NCT06271070
Title: Analysis of Correlation Between Skin Carotenoid Level and Basic Indicators of Health Status Related to Lifestyle in Vietnamese: An Observational Study
Status: Completed | Type: Observational
Sponsor: KAGOME CO., LTD. (Industry)
Responsible Party: Sponsor
Other Study IDs: 2023-R23
Record Dates: First submitted 2024-01-30; First posted 2024-02-21 (Actual); Last update posted 2025-04-16 (Actual); Status verified 2025-04

CONDITIONS: Lifestyle Risk Reduction
MeSH Terms: conditions — Risk Reduction Behavior

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

INTERVENTIONS:
Other: Non-intervention — Non

SUMMARY:
To clarify the relationship between vegetable intake and lifestyle-related disease in Vietnam, we measure skin carotenoid levels and basic indicators of health status related to lifestyle and analyze the correlation between them. This is an important study that can lead to dietary suggestions for preventing lifestyle-related diseases in Vietnam.

ELIGIBILITY:
Inclusion Criteria:

1. Adults aged 18 years or older
2. Healthy people or patients with metabolic diseases as obesity, diabetes, hypertension, lipid abnormalities, hyperuricemia
3. People who agreed to participate in the study and be able to complete the Informed Consent Form

Exclusion Criteria:

1. Hospitalized patients
2. Patients with other diseases than metabolic diseases as written in inclusion criteria.
3. People judged to be inappropriate by the principal investigator

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Visitors to Dr. Binh_TeleClinic
Sampling Method: Non-Probability Sample
Enrollment: 300 (Actual)
Dates: Start 2024-01-30 (Actual); Primary Completion 2024-05-31 (Actual); Study Completion 2024-12-31 (Actual)

PRIMARY OUTCOMES:
Skin carotenoid level | single day
Blood markers of lifestyle-related diseases | single day
  Blood glucose level, Blood lipid (triglyceride, HDL-cholesterol, LDL-cholesterol) levels
BMI | single day
Body fat percentage | single day
Blood pressure | single day

SECONDARY OUTCOMES:
Questionnaire | single day
  Gender, Age, Income (optional-if subject agree), Academic background, Medication, Diet therapy, Lifestyle behavior (Smoking, Drinking, Vegetable intake)

CONTACTS AND LOCATIONS:
Overall Officials: Nguyen Thuy Lan, Doctor, Principal Investigator — Dr. Binh_Teleclinic - Branch of E2E Solution Company Limited
Locations (1):
- Dr. Binh_Teleclinic - Branch of E2E Solution Company Limited, Hanoi, Vietnam

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Matsumoto M, Suganuma H, Shimizu S, Hayashi H, Sawada K, Tokuda I, Ihara K, Nakaji S. Skin Carotenoid Level as an Alternative Marker of Serum Total Carotenoid Concentration and Vegetable Intake Correlates with Biomarkers of Circulatory Diseases and Metabolic Syndrome. Nutrients. 2020 Jun 19;12(6):1825. doi: 10.3390/nu12061825. PMID 32575348
- [Derived] Yoshida K, Nakazawa Y, Nguyen TL, Nguyen DH, Anh CX, Takahashi S, Suzuki S, Binh VQ. Higher skin carotenoid levels are associated with lower risks of metabolic syndrome: a cross-sectional study in Vietnamese participants. Front Nutr. 2026 Jan 22;12:1715158. doi: 10.3389/fnut.2025.1715158. eCollection 2025. PMID 41659800